CLINICAL TRIAL: NCT02415400
Title: An Open-label, 2 x 2 Factorial, Randomized Controlled, Clinical Trial to Evaluate the Safety of Apixaban vs. Vitamin K Antagonist and Aspirin vs. Aspirin Placebo in Patients With Atrial Fibrillation and Acute Coronary Syndrome or Percutaneous Coronary Intervention
Brief Title: A Study of Apixaban in Patients With Atrial Fibrillation, Not Caused by a Heart Valve Problem, Who Are at Risk for Thrombosis (Blood Clots) Due to Having Had a Recent Coronary Event, Such as a Heart Attack or a Procedure to Open the Vessels of the Heart
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry); Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: CV185-316; 2014-002004-24 (EudraCT Number)
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Results first posted 2020-02-07 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Acute Coronary Syndromes
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — apixaban; acarboxyprothrombin; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Apixaban (Active Comparator): 5 mg or 2.5 mg Apixaban tablets orally twice per day
  Interventions: Drug: Apixaban
- Vitamin K Antagonist (Active Comparator): VKA tablets orally once daily
  Interventions: Drug: vitamin K antagonist
- Acetylsalicylic acid film coated tablet (Placebo Comparator): 81 mg Acetylsalicylic acid film coated tablet orally once daily
  Interventions: Drug: Acetylsalicylic acid
- Placebo matching Acetylsalicylic acid film coated tablet (Placebo Comparator): Placebo matching Acetylsalicylic acid film coated tablet once daily
  Interventions: Other: Acetylsalicylic acid placebo

INTERVENTIONS:
Drug: Apixaban
  Other Names: BMS-562247
  Arms: Apixaban
Drug: vitamin K antagonist
  Arms: Vitamin K Antagonist
Drug: Acetylsalicylic acid
  Other Names: Aspirin 81 mg
  Arms: Acetylsalicylic acid film coated tablet
Other: Acetylsalicylic acid placebo
  Other Names: aspirin placebo
  Arms: Placebo matching Acetylsalicylic acid film coated tablet

SUMMARY:
The purpose of this study is to determine if Apixaban is safer than a Vitamin K Antagonist given for 6 months in terms of bleeding in patients with an irregular heart beat (atrial fibrillation) and a recent heart attack or a recent procedure to open up a blood vessel in the heart. All patients would also be taking a class of medicines called P2Y12 inhibitors (such as clopidogrel/Plavix) and be treated for up to 6 months. The primary focus will be a comparison of the bleeding risk of Apixaban, with or without aspirin, versus a Vitamin K antagonist, such as warfarin, with or without aspirin.

DETAILED DESCRIPTION:
Patients will be recruited from either inpatient coronary care or general medical units, or recruited from outpatient cardiology offices.

Masking:

Apixaban: Open label.

VKA: Open label.

Acetylsalicylic acid film coated tablet: Double Blinded.

Placebo matching Acetylsalicylic acid film coated tablet: Double Blinded.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Adults with either active or a history of non-valvular atrial fibrillation or flutter with the planned or existing use of an oral anticoagulant for prophylaxis of thromboembolism. In addition, subjects must have had an acute coronary syndrome or percutaneous coronary intervention with a stent within the prior 14 days
* Planned use of antiplatelet agents for at least 1 to 6 months
* Males and Females ≥ 18 years of age
* Women of childbearing potential must have a negative serum or urine pregnancy test within 24 hours prior to the start of study drug

Exclusion Criteria:

* Conditions other than atrial fibrillation that require chronic anticoagulation. (e.g. prosthetic mechanical heart valve)
* Severe renal insufficiency (serum creatinine > 2.5 mg/dL or a calculated creatinine clearance < 30 mL/min
* Patients with a history of intracranial hemorrhage
* Patients have had or will undergo Coronary arterial bypass graft (CABG) for their index acute coronary syndrome (ACS) event
* Patients with known ongoing bleeding and patients with known coagulopathies
* Any contraindications or allergies to VKA, apixaban, or to intended P2Y12 antagonists or to aspirin

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4614 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2018-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (509):
- United States (140):
  - Cardiovascular Associates of the Southeast, LLC, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Heart Rhythm Center, Phoenix, Arizona
  - Local Institution, Phoenix, Arizona
  - Scottsdale Osborn Medical Center, Scottsdale, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Phoenix, Arkansas
  - Comprehensive Cardiovascular Specialists, Alhambra, California
  - Local Institution, Culver City, California
  - Washington Township Medical Foundation, Fremont, California
  - California Heart Specialist, Inc., Huntington Beach, California
  - Foundation For Cardiovascular Medicine, La Jolla, California
  - Local Institution, Long Beach, California
  - Local Institution, Rancho Mirage, California
  - Local Institution, San Diego, California
  - Manshadi Heart Institute, Stockton, California
  - Local Institution, Torrance, California
  - University Of Colorado, Aurora, Colorado
  - Colorado Heart and Vascular, Lakewood, Colorado
  - Local Institution, Norwalk, Connecticut
  - Local Institution, Wilmington, Delaware
  - Orlando Heart Specialists, Altamonte Springs, Florida
  - Local Institution, Bradenton, Florida
  - Clearwater Cardiovascular and Interventional Consultants, Clearwater, Florida
  - Local Institution, Clearwater, Florida
  - Daytona Heart Group, Daytona Beach, Florida
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Jacksonville Beach, Florida
  - Tenet Florida Physician Services, Jupiter, Florida
  - Local Institution, Lake Mary, Florida
  - Local Institution, Miami, Florida
  - Mediquest Research, Ocala, Florida
  - Local Institution, Orlando, Florida
  - CP Cardiology Partners, Palm Beach Gardens, Florida
  - Bayfront Health St. Petersburg, St. Petersburg, Florida
  - Local Institution, Tampa, Florida
  - Cardiology Partners, Wellington, Florida
  - Athens Regional Cariology Group, Athens, Georgia
  - Local Institution, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Georgia Heart Specialists, Covington, Georgia
  - Local Institution, Cumming, Georgia
  - Local Institution, Tucker, Georgia
  - Saint Lukes Idaho Cardiology Associates, Boise, Idaho
  - Medicoricium, LLC, Fairview Heights, Illinois
  - Gateway Cardiology PC, Jerseyville, Illinois
  - Advocate Medical Group ? Cardiology and Pulmonology, Normal, Illinois
  - South Suburban Cardiology, Olympia Fields, Illinois
  - Local Institution, Bloomington, Indiana
  - Elkhart Clinic LLC, Elkhart, Indiana
  - Roudebush VA Medical Center, Indianapolis, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - Northeast Iowa Family Practice Center, Waterloo, Iowa
  - Local Institution, Kansas City, Kansas
  - Local Institution, Wichita, Kansas
  - Saint Elizabeth Healthcare, Crestview Hills, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Alexandria Cardiology Clinic, Alexandria, Louisiana
  - Imperial Health, Lake Charles, Louisiana
  - Local Institution, Minden, Louisiana
  - Clinical Trials of America LA LLC - PPDS, Monroe, Louisiana
  - Local Institution, Natick, Massachusetts
  - Great Lakes Heart Center of Alpena, Alpena, Michigan
  - Local Institution, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Local Institution, Detroit, Michigan
  - Local Institution, Lansing, Michigan
  - Covenant Center for the Heart, Saginaw, Michigan
  - Metropolitan Cardiology Consultants, Minneapolis, Minnesota
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Local Institution, Jackson, Mississippi
  - Cardiology Associates Research LLC, Tupelo, Mississippi
  - Missouri Cardiovascular Specialists, Columbia, Missouri
  - Local Institution, Columbia, Missouri
  - Freeman Health System, Joplin, Missouri
  - Cox Health Systems, Springfield, Missouri
  - Gateway Cardiology PC, St Louis, Missouri
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Local Institution, Billings, Montana
  - Bryan Heart Hospital, Lincoln, Nebraska
  - HCP Clinical Research LLC, Las Vegas, Nevada
  - Renown Regional Medical Center., Reno, Nevada
  - New Jersey Heart, Linden, New Jersey
  - Capital Cardiology Associates, Albany, New York
  - New York-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Local Institution, Brooklyn, New York
  - Buffalo Heart Group LLP, Buffalo, New York
  - Mount Sinai-St. Lukes, New York, New York
  - Hudson Valley Cardiovascular Practice, PC, Poughkeepsie, New York
  - Asheville Cardiology Associates PA, Asheville, North Carolina
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Clinical Trials of America-NC, LLC - PPDS, Lenoir, North Carolina
  - Duke Cardiology and Cardiovascular Surgery of Lumberton, Lumberton, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Aultman Hospital, Canton, Ohio
  - Local Institution, Columbus, Ohio
  - Local Institution, Kettering, Ohio
  - Local Institution, Willoughby, Ohio
  - Saint Vincent Hospital, Erie, Pennsylvania
  - Heart Group, Lancaster, Pennsylvania
  - Mercer Bucks Cardiology, Newton, Pennsylvania
  - WellSpan York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Columbia Heart, Columbia, South Carolina
  - Upstate Cardiology PA, Greenville, South Carolina
  - Roper St. Francis Healthcare, North Charleston, South Carolina
  - Carolina Cardiology Clinical Research Institute, Rock Hill, South Carolina
  - Local Institution, Germantown, Tennessee
  - Research Associates of Jackson, Jackson, Tennessee
  - Cardiovascular Research of Knoxville, Knoxville, Tennessee
  - Knoxville Health Managment Associates Cardiology PPM LLC, Knoxville, Tennessee
  - Parkway Cardiology Associates PC, Oak Ridge, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, Dallas, Texas
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - Angiocardiac Care of Texas PA, Houston, Texas
  - Local Institution, Houston, Texas
  - Grace Research, LLC, Huntsville, Texas
  - Local Institution, Huntsville, Texas
  - Local Institution, Katy, Texas
  - Caprock Cardiac Center Research Institute, Lubbock, Texas
  - Local Institution, Plano, Texas
  - Local Institution, San Antonio, Texas
  - Mercury Medical LLC, San Antonio, Texas
  - Local Institution, Sealy, Texas
  - Local Institution, Sugar Land, Texas
  - Victoria Heart and Vascular Center, Victoria, Texas
  - University of Vermont, Burlington, Vermont
  - Virginia Heart, Falls Church, Virginia
  - Virginia Heart Group Ltd, Leesburg, Virginia
  - CJW Medical Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - St Mary's Medical Center, Huntington, West Virginia
  - Aspirus Research Institute, Wausau, Wisconsin
- Argentina (19):
  - Local Institution, Buenos Aires, BUA
  - Local Institution, Bahía Blanca, Buenos Aires
  - Local Institution, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution, Coronel Suárez, Buenos Aires
  - Local Institution, Lanús Oeste, Buenos Aires
  - Local Institution, Mar del Plata, Buenos Aires
  - Local Institution, Quilmes, Buenos Aires
  - Local Institution, Ramos Mejía, Buenos Aires
  - Local Institution, Vicente López, Buenos Aires
  - Local Institution, Resistencia, Chaco Province
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Villa Allende, Córdoba Province
  - Local Institution, Villa María, Córdoba Province
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, Buenos Aires
  - Local Institution, Corrientes
  - Local Institution, Córdoba
  - Local Institution, Santa Fe
  - Local Institution, Santiago del Estero
- Australia (5):
  - Local Institution, Concord, New South Wales
  - Local Institution, Port Macquarie, New South Wales
  - Local Institution, Milton, Queensland
  - Local Institution, Elizabeth Vale, South Australia
  - Local Institution, Bedford Park
- Austria (3):
  - Local Institution, Graz
  - Local Institution, Linz
  - Local Institution, Vienna
- Belgium (10):
  - Local Institution, Aalst
  - Local Institution, Antwerp
  - Local Institution, Bonheiden
  - Local Institution, Brasschaat
  - Local Institution, Brussels
  - Local Institution, Ghent
  - Local Institution, Ieper
  - Local Institution, Leuven
  - Local Institution, Wilrijk
  - Local Institution, Yvoir
- Brazil (26):
  - Local Institution, Colatina, Espírito Santo
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Brasília, Federal District
  - Local Institution, Aparecida de Goiânia, Goiás
  - Local Institution, Goiânia, Goiás
  - Local Institution, Belo Horizonte, Minas Gerais
  - Local Institution, Uberaba, Minas Gerais
  - Local Institution, Uberlândia, Minas Gerais
  - Local Institution, Campina Grande do Sul, Paraná
  - Local Institution, Londrina, Paraná
  - Local Institution, Belém, Pará
  - Local Institution, Recife, Pernambuco
  - Local Institution, Canoas, Rio Grande do Sul
  - Local Institution, Passo Fundo, Rio Grande do Sul
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Blumenau, Santa Catarina
  - Local Institution, Itajaí, Santa Catarina
  - Local Institution, Campinas, São Paulo
  - Local Institution, Limeira, São Paulo
  - Local Institution, Marília, São Paulo
  - Local Institution, S?o Paulo, São Paulo
  - Local Institution, Santo André, São Paulo
  - Local Institution, São José do Rio Preto, São Paulo
  - Local Institution, Votuporanga, São Paulo
  - Local Institution, Rio de Janeiro
  - Local Institution, São Paulo
- Bulgaria (12):
  - Local Institution, Burgas
  - Local Institution, Dimitrovgrad
  - Local Institution, Haskovo
  - Local Institution, Montana
  - Local Institution, Pazardzhik
  - Local Institution, Pleven
  - Local Institution, Plovdiv
  - Local Institution, Sandanski
  - Local Institution, Smolyan
  - Local Institution, Sofia
  - Local Institution, Veliko Tarnova
  - Local Institution, Vidin
- Canada (22):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Kelowna, British Columbia
  - Local Institution, New Westminster, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Winnepeg, Manitoba
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Cambridge, Ontario
  - Local Institution, Greater Sudbury, Ontario
  - Local Institution, London, Ontario
  - Local Institution, Oshawa, Ontario
  - Local Institution, Scarborough Village, Ontario
  - Local Institution, Waterloo, Ontario
  - Local Institution, Green Field Park, Quebec
  - Local Institution, Laval, Quebec
  - Local Institution, Longueuil, Quebec
  - Local Institution, Montreal, Quebec
  - Local Institution, Saint-Jean-sur-Richelieu, Quebec
  - Local Institution, Saint-Jérôme, Quebec
  - Local Institution, Sherbrooke, Quebec
  - Local Institution, St-Georges, Beauce, Quebec
  - Local Institution, Regina, Saskatchewan
  - Local Institution, Montreal
- Local Institution, Santiago, Santiago Metropolitan, Chile
- Colombia (5):
  - Local Institution, Barranquilla
  - Local Institution, Bogotá
  - Local Institution, Cali
  - Local Institution, Espinal
  - Local Institution, Medellín
- Croatia (13):
  - Local Institution, Čakovec
  - Local Institution, Dubrovnik
  - Local Institution, Karlovac
  - Local Institution, Krapinske Toplice
  - Local Institution, Opatija
  - Local Institution, Osijek
  - Local Institution, Rijeka
  - Local Institution, Slavonski Brod
  - Local Institution, Šibenik
  - Local Institution, Virovitica
  - Local Institution, Zabok
  - Local Institution, Zadar
  - Local Institution, Zagreb
- Czechia (4):
  - Local Institution, Prague
  - Local Institution, Tábor
  - Local Institution, Ústí nad Orlicí
  - Local Institution, Zlín
- Denmark (11):
  - Local Institution, Aabenraa
  - Local Institution, Aarhus
  - Local Institution, Copenhagen
  - Local Institution, Frederiksburg
  - Local Institution, Hellerup
  - Local Institution, Hillerød
  - Local Institution, Holb?k
  - Local Institution, Hvidovre
  - Local Institution, Randers
  - Local Institution, Roskilde
  - Local Institution, Slagelse
- France (10):
  - Local Institution, Besançon
  - Local Institution, Caen
  - Local Institution, Chambray-lès-Tours
  - Local Institution, Le Coudray
  - Local Institution, Lyon
  - Local Institution, Marseille
  - Local Institution, Nîmes
  - Local Institution, Pau
  - Local Institution, Pessac
  - Local Institution, Toulouse
- Germany (43):
  - Local Institution, Bad Friedrichshall
  - Local Institution, Bad Homburg
  - Local Institution, Berlin
  - Local Institution, Bielefeld
  - Local Institution, Brandenburg
  - Local Institution, Bremen
  - Local Institution, Chemnitz
  - Local Institution, Cologne
  - Local Institution, Dortmund
  - Local Institution, Dresden
  - Local Institution, Erfurt
  - Local Institution, Erlangen
  - Local Institution, Essen
  - Local Institution, Frankfurt am Main
  - Local Institution, Freiburg im Breisgau
  - Local Institution, Göttingen
  - Local Institution, Greifswald
  - Local Institution, Hamburg
  - Local Institution, Hennigsdorf
  - Local Institution, Hoyerswerda
  - Local Institution, Jena
  - Local Institution, Karlsbad
  - Local Institution, Kassel
  - Local Institution, Lahr
  - Local Institution, Leipzig
  - Local Institution, Limburg
  - Local Institution, Lübeck
  - Local Institution, Lüdenscheid
  - Local Institution, Magdeburg
  - Local Institution, Mainz
  - Local Institution, Mannheim
  - Local Institution, Neuss
  - Local Institution, Papenburg
  - Local Institution, Regensburg
  - Local Institution, Rostock
  - Local Institution, Stendal
  - Local Institution, Straubing
  - Local Institution, Tübingen
  - Local Institution, Ulm
  - Local Institution, Villingen-Schwenningen
  - Local Institution, Weiden i.d.OPf.
  - Local Institution, Worms
  - Local Institution, Würzburg
- Hungary (9):
  - Local Institution, Baja, Bács-Kiskun county
  - Local Institution, Békéscsaba
  - Local Institution, Budapest
  - Local Institution, Keszthely
  - Local Institution, Mosonmagyaróvár
  - Local Institution, Pécs
  - Local Institution, Szeged
  - Local Institution, Szekszárd
  - Local Institution, Szolnok
- India (12):
  - Local Institution, Ahmedabad, Gujarat
  - Local Institution, Bangalore, Karnataka
  - Local Institution, Amritsar
  - Local Institution, Jaipur
  - Local Institution, Lucknow
  - Local Institution, Madurai
  - Local Institution, Mangalore
  - Local Institution, New Delhi
  - Local Institution, Noida
  - Local Institution, Shivamogga
  - Local Institution, Vadodara
  - Local Institution, Vijayawada
- Israel (12):
  - Local Institution, Afula
  - Local Institution, Ashkelon
  - Local Institution, Hadera
  - Local Institution, Haifa
  - Local Institution, Herzliya
  - Local Institution, Holon
  - Local Institution, Jerusalem
  - Local Institution, Ramat Gan
  - Local Institution, Rehovot
  - Local Institution, Safed
  - Local Institution, Tel Aviv
  - Local Institution, Tiberias
- Local Institution, Grosseto, Italy
- Mexico (13):
  - Local Institution, Torreón, Coahuila
  - Local Institution, León, Guanajuato
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Querétaro City, Querétaro
  - Local Institution, San Juan del Río, Querétaro
  - Local Institution, Culiacán, Sinaloa
  - Local Institution, Aguascalientes
  - Local Institution, Durango
  - Local Institution, Puebla City
  - Local Institution, San Luis Potosí City
  - Local Institution, Tlalnepantla
  - Local Institution, Veracruz
- Netherlands (11):
  - Local Institution, Amsterdam
  - Local Institution, Arnhem
  - Local Institution, Breda
  - Local Institution, Ede
  - Local Institution, Groningen
  - Local Institution, Hardenberg
  - Local Institution, Maastricht
  - Local Institution, Nieuwegein
  - Local Institution, Rotterdam
  - Local Institution, Tilburg
  - Local Institution, Uden
- Norway (5):
  - Local Institution, Bod?
  - Local Institution, Oslo
  - Local Institution, Skien
  - Local Institution, Stavanger
  - Local Institution, Tromsø
- Peru (4):
  - Local Institution, Miraflores, Lima region
  - Local Institution, Callao
  - Local Institution, Cusco
  - Local Institution, Lima
- Poland (18):
  - Local Institution, Poznan, Greater Poland Voivodeship
  - Local Institution, Bialystok
  - Local Institution, Bydgoszcz
  - Local Institution, Bytom
  - Local Institution, Chojnice
  - Local Institution, Gdynia
  - Local Institution, Katowice
  - Local Institution, Kielce
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Lubin
  - Local Institution, Opole
  - Local Institution, Płock
  - Local Institution, Siemianowice Śląskie
  - Local Institution, Torun
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
  - Local Institution, Włocławek
- Portugal (10):
  - Local Institution, Almada
  - Local Institution, Aveiro
  - Local Institution, Braga
  - Local Institution, Coimbra
  - Local Institution, Covilha
  - Local Institution, Guimar?es
  - Local Institution, Leiria
  - Local Institution, Lisbon
  - Local Institution, Senhora de Hora, Matosinhos
  - Local Institution, Vila Real
- Local Institution, Caguas, Puerto Rico
- Romania (11):
  - Local Institution, Baia Mare
  - Local Institution, Brasov
  - Local Institution, Bucharest
  - Local Institution, Cluj-Napoca
  - Local Institution, Craiova
  - Local Institution, Oradea
  - Local Institution, Piteşti
  - Local Institution, Sibiu
  - Local Institution, Târgovişte
  - Local Institution, Târgu Mureş
  - Local Institution, Timișoara
- Russia (11):
  - Local Institution, Gatchina
  - Local Institution, Kazan'
  - Local Institution, Krasnodar
  - Local Institution, Moscow
  - Local Institution, Novosibirsk
  - Local Institution, Saint Petersburg
  - Local Institution, Samara
  - Local Institution, Saratov
  - Local Institution, Sochi
  - Local Institution, Tyumen
  - Local Institution, Yekaterinburg
- Serbia (5):
  - Local Institution, Belgarde
  - Local Institution, Belgrade
  - Local Institution, Kamenitz
  - Local Institution, Niš
  - Local Institution, Užice
- Slovakia (9):
  - Local Institution, Banská Bystrica
  - Local Institution, Bardejov
  - Local Institution, Bratislava
  - Local Institution, Brezno
  - Local Institution, Košice
  - Local Institution, Nitra
  - Local Institution, Spišská Nová Ves
  - Local Institution, Trebišov
  - Local Institution, Trenčín
- South Korea (8):
  - Local Institution, Busan
  - Local Institution, Changwon
  - Local Institution, Daegu
  - Local Institution, Daejeon
  - Local Institution, Gwangju
  - Local Institution, Incheon
  - Local Institution, Seongnam-si
  - Local Institution, Seoul
- Spain (11):
  - Local Institution, Majadahonda, Madrid
  - Local Institution, Alicante
  - Local Institution, Barcelona
  - Local Institution, Córdoba
  - Local Institution, Donostia / San Sebastian
  - Local Institution, Huelva
  - Local Institution, Madrid
  - Local Institution, Marbella
  - Local Institution, Málaga
  - Local Institution, Palma de Mallorca
  - Local Institution, Valencia
- Sweden (7):
  - Local Institution, Eskilstuna
  - Local Institution, Gothenburg
  - Local Institution, Jönköping
  - Local Institution, Östersund
  - Local Institution, Skellefteå
  - Local Institution, Stockholm
  - Local Institution, Uppsala
- Switzerland (3):
  - Local Institution, Bern
  - Local Institution, Geneva
  - Local Institution, Winterthur
- Ukraine (12):
  - Local Institution, Cherkasy
  - Local Institution, Chernivtsi
  - Local Institution, Dnipropetrovsk
  - Local Institution, Ivano-Frankivsk
  - Local Institution, Kharkiv
  - Local Institution, Kyiv
  - Local Institution, Lutsk
  - Local Institution, Mykolaiv
  - Local Institution, Odesa
  - Local Institution, Uzhhorod
  - Local Institution, Vinnytsia
  - Local Institution, Zhaporizhzhya
- United Kingdom (11):
  - Local Institution, Bournemouth, Dorset
  - Local Institution, Kirkcaldy, FIFE
  - Local Institution, Stevenage, Hertfordshire
  - Local Institution, Liverpool, Merseyside
  - Local Institution, Northampton, Northamptonshire
  - Local Institution, Doncaster, South Yorkshire
  - Local Institution, Sheffield, South Yorkshire
  - Local Institution, Birmingham
  - Local Institution, Dudley, West Midlands
  - Local Institution, Dundee
  - Local Institution, Wolverhampton
- Local Institution, Christiansted, Virgin Islands

REFERENCES:
- [Derived] Fudim M, Lopes RD, Wojdyla DM, Mehran R, Khan MS, Granger CB, Goodman SG, Aronson R, Windecker S, Alexander JH. Apixaban Dose in Patients With Atrial Fibrillation and Acute Coronary Syndrome and/or Undergoing Percutaneous Coronary Intervention: Insights From AUGUSTUS. JACC Adv. 2025 Apr;4(4):101665. doi: 10.1016/j.jacadv.2025.101665. Epub 2025 Mar 20. PMID 40117694
- [Derived] Tannu M, Lopes RD, Wojdyla DM, Goodman SG, Aronson R, Mehran R, Granger CB, Windecker S, Alexander JH, Jones WS. Antithrombotic Therapy to Minimize Total Events After ACS or PCI in Atrial Fibrillation: Insights From AUGUSTUS. J Am Coll Cardiol. 2025 Mar 25;85(11):1157-1168. doi: 10.1016/j.jacc.2024.10.125. Epub 2025 Feb 5. PMID 39918467
- [Derived] Fanaroff AC, Vora AN, Wojdyla DM, Mehran R, Granger CB, Goodman SG, Aronson R, Windecker S, Alexander JH, Lopes RD. Effect of apixaban versus vitamin K antagonist and aspirin versus placebo on days alive and out of hospital: An analysis from AUGUSTUS. Am Heart J. 2025 Feb;280:60-69. doi: 10.1016/j.ahj.2024.11.005. Epub 2024 Nov 17. PMID 39557109
- [Derived] Fanaroff AC, Wojdyla DM, Granger CB, Goodman SG, Aronson RS, Windecker S, Mehran R, Alexander JH, Lopes RD. Relative Benefit of Dual Versus Single Antiplatelet Therapy Among Patients With Atrial Fibrillation on Oral Anticoagulation According to Time After ACS and PCI: Insights From the AUGUSTUS Trial. Circ Cardiovasc Interv. 2024 Nov;17(11):e013596. doi: 10.1161/CIRCINTERVENTIONS.123.013596. Epub 2024 Nov 6. PMID 39502066
- [Derived] Berwanger O, Wojdyla DM, Fanaroff AC, Budaj A, Granger CB, Mehran R, Aronson R, Windecker S, Goodman SG, Alexander JH, Lopes RD. Antithrombotic Strategies in Atrial Fibrillation After ACS and/or PCI: A 4-Way Comparison From AUGUSTUS. J Am Coll Cardiol. 2024 Sep 3;84(10):875-885. doi: 10.1016/j.jacc.2024.06.022. PMID 39197976
- [Derived] Guimaraes PO, Lopes RD, Wojdyla DM, Alexander JH, Goodman SG, Aronson R, Halvorsen S, Sinnaeve P, Vinereanu D, Storey RF, Berwanger O, Windecker S, Mehran R, Granger CB, Alexander KP; AUGUSTUS Investigators. Antithrombotic Strategies According to Age: Insights from the AUGUSTUS Trial. Am J Med. 2024 Oct;137(10):958-965. doi: 10.1016/j.amjmed.2024.06.001. Epub 2024 Jun 13. PMID 38876331
- [Derived] Bahit MC, Vora AN, Li Z, Wojdyla DM, Thomas L, Goodman SG, Aronson R, Jordan JD, Kolls BJ, Dombrowski KE, Vinereanu D, Halvorsen S, Berwanger O, Windecker S, Mehran R, Granger CB, Alexander JH, Lopes RD. Apixaban or Warfarin and Aspirin or Placebo After Acute Coronary Syndrome or Percutaneous Coronary Intervention in Patients With Atrial Fibrillation and Prior Stroke: A Post Hoc Analysis From the AUGUSTUS Trial. JAMA Cardiol. 2022 Jul 1;7(7):682-689. doi: 10.1001/jamacardio.2022.1166. PMID 35612866
- [Derived] Welsh RC, Dehghani P, Lopes R, Wojdyla DM, Aronson R, Granger CB, Windecker S, Vora AN, Vinereanu D, Halvorsen S, Parkhomenko A, Mehran R, Alexander JH, Goodman S. Impact of prior oral anticoagulant use and outcomes on patients from secondary analysis in the AUGUSTUS trial. Open Heart. 2022 Feb;9(1):e001892. doi: 10.1136/openhrt-2021-001892. PMID 35172988
- [Derived] Harskamp RE, Fanaroff AC, Lopes RD, Wojdyla DM, Goodman SG, Thomas LE, Aronson R, Windecker S, Mehran R, Granger CB, Alexander JH. Antithrombotic Therapy in Patients With Atrial Fibrillation After Acute Coronary Syndromes or Percutaneous Intervention. J Am Coll Cardiol. 2022 Feb 8;79(5):417-427. doi: 10.1016/j.jacc.2021.11.035. PMID 35115097
- [Derived] Hijazi Z, Alexander JH, Li Z, Wojdyla DM, Mehran R, Granger CB, Parkhomenko A, Bahit MC, Windecker S, Aronson R, Berwanger O, Halvorsen S, de Waha-Thiele S, Sinnaeve P, Darius H, Storey RF, Lopes RD. Apixaban or Vitamin K Antagonists and Aspirin or Placebo According to Kidney Function in Patients With Atrial Fibrillation After Acute Coronary Syndrome or Percutaneous Coronary Intervention: Insights From the AUGUSTUS Trial. Circulation. 2021 Mar 23;143(12):1215-1223. doi: 10.1161/CIRCULATIONAHA.120.051020. Epub 2021 Jan 19. PMID 33461308
- [Derived] Alexander JH, Wojdyla D, Vora AN, Thomas L, Granger CB, Goodman SG, Aronson R, Windecker S, Mehran R, Lopes RD. Risk/Benefit Tradeoff of Antithrombotic Therapy in Patients With Atrial Fibrillation Early and Late After an Acute Coronary Syndrome or Percutaneous Coronary Intervention: Insights From AUGUSTUS. Circulation. 2020 May 19;141(20):1618-1627. doi: 10.1161/CIRCULATIONAHA.120.046534. Epub 2020 Mar 29. PMID 32223444
- [Derived] Lopes RD, Leonardi S, Wojdyla DM, Vora AN, Thomas L, Storey RF, Vinereanu D, Granger CB, Goodman SG, Aronson R, Windecker S, Thiele H, Valgimigli M, Mehran R, Alexander JH. Stent Thrombosis in Patients With Atrial Fibrillation Undergoing Coronary Stenting in the AUGUSTUS Trial. Circulation. 2020 Mar 3;141(9):781-783. doi: 10.1161/CIRCULATIONAHA.119.044584. Epub 2019 Nov 11. No abstract available. PMID 31707833
- [Derived] Windecker S, Lopes RD, Massaro T, Jones-Burton C, Granger CB, Aronson R, Heizer G, Goodman SG, Darius H, Jones WS, Aschermann M, Brieger D, Cura F, Engstrom T, Fridrich V, Halvorsen S, Huber K, Kang HJ, Leiva-Pons JL, Lewis BS, Malaga G, Meneveau N, Merkely B, Milicic D, Morais J, Potpara TS, Raev D, Sabate M, de Waha-Thiele S, Welsh RC, Xavier D, Mehran R, Alexander JH; AUGUSTUS Investigators. Antithrombotic Therapy in Patients With Atrial Fibrillation and Acute Coronary Syndrome Treated Medically or With Percutaneous Coronary Intervention or Undergoing Elective Percutaneous Coronary Intervention: Insights From the AUGUSTUS Trial. Circulation. 2019 Dec 3;140(23):1921-1932. doi: 10.1161/CIRCULATIONAHA.119.043308. Epub 2019 Sep 26. PMID 31557056
- [Derived] Lopes RD, Heizer G, Aronson R, Vora AN, Massaro T, Mehran R, Goodman SG, Windecker S, Darius H, Li J, Averkov O, Bahit MC, Berwanger O, Budaj A, Hijazi Z, Parkhomenko A, Sinnaeve P, Storey RF, Thiele H, Vinereanu D, Granger CB, Alexander JH; AUGUSTUS Investigators. Antithrombotic Therapy after Acute Coronary Syndrome or PCI in Atrial Fibrillation. N Engl J Med. 2019 Apr 18;380(16):1509-1524. doi: 10.1056/NEJMoa1817083. Epub 2019 Mar 17. PMID 30883055
- [Derived] Lopes RD, Vora AN, Liaw D, Granger CB, Darius H, Goodman SG, Mehran R, Windecker S, Alexander JH. An open-Label, 2 x 2 factorial, randomized controlled trial to evaluate the safety of apixaban vs. vitamin K antagonist and aspirin vs. placebo in patients with atrial fibrillation and acute coronary syndrome and/or percutaneous coronary intervention: Rationale and design of the AUGUSTUS trial. Am Heart J. 2018 Jun;200:17-23. doi: 10.1016/j.ahj.2018.03.001. Epub 2018 Mar 9. PMID 29898844
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4683 participants enrolled, 4614 randomized. Reasons not randomized: 2 adverse event; 1 request to stop therapy; 12 withdrew consent; 1 lost to follow-up; 1 poor/non-compliance; 35 no longer met criteria; 2 admin reasons by Sponsor; 10 lack of IP at site; 1 IWRS down; 2 physician recommended; 1 leaving the country; 1 pharmacogenetic sample positive
Groups:
- Apixaban With Acetylsalicylic Acid Film Coated Tablet: 5 mg or 2.5 mg Apixaban tablets orally twice per day with 81 mg Acetylsalicylic acid film coated tablet orally once daily with concomitant P2Y12 inhibitor therapy
- Apixaban With Placebo Matching Acetylsalicylic Acid: 5 mg or 2.5 mg Apixaban tablets orally twice per day with placebo matching Acetylsalicylic acid film coated tablet orally once daily with concomitant P2Y12 inhibitor therapy
- Vitamin K Antagonist (VKA) With Acetylsalicylic Acid: VKA tablets orally once daily with 81 mg Acetylsalicylic acid film coated tablet orally once daily with concomitant P2Y12 inhibitor therapy
- VKA With Placebo Matching Acetylsalicylic Acid: VKA tablets orally once daily with placebo matching Acetylsalicylic acid film coated tablet orally once daily with concomitant P2Y12 inhibitor therapy
Period: Overall Study
Arm/Group | Apixaban With Acetylsalicylic Acid Film Coated Tablet | Apixaban With Placebo Matching Acetylsalicylic Acid | Vitamin K Antagonist (VKA) With Acetylsalicylic Acid | VKA With Placebo Matching Acetylsalicylic Acid
Started (Started = Randomized) | 1153 | 1153 | 1154 | 1154
Completed (Completed = Completing the period) | 1087 | 1091 | 1069 | 1071
Not Completed | 66 | 62 | 85 | 83
Not completed — Adverse Event | 0 | 1 | 1 | 2
Not completed — Participant request to stop therapy | 4 | 3 | 8 | 6
Not completed — Participant withdrew consent | 14 | 12 | 30 | 21
Not completed — Death | 39 | 41 | 35 | 42
Not completed — Lost to Follow-up | 3 | 3 | 2 | 5
Not completed — Poor/Non-Compliance | 0 | 1 | 3 | 4
Not completed — Participant no longer meets criteria | 2 | 0 | 0 | 1
Not completed — Participant doesn't answer phone | 1 | 0 | 0 | 0
Not completed — Participant wanted home visits | 1 | 0 | 0 | 0
Not completed — Randomized in error | 2 | 0 | 0 | 0
Not completed — No study drug on site | 0 | 1 | 0 | 0
Not completed — Stroke and stroke rehabilitation | 0 | 0 | 1 | 0
Not completed — Coagulation values cannot be set | 0 | 0 | 1 | 0
Not completed — State regulations prevent participation | 0 | 0 | 1 | 0
Not completed — Poor treatment monitoring | 0 | 0 | 1 | 0
Not completed — Participant in jail | 0 | 0 | 1 | 0
Not completed — Investigator decision | 0 | 0 | 1 | 1
Not completed — Site closure; participant won't transfer | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Vitamin K Antagonist (VKA) With Acetylsalicylic: VKA tablets orally once daily with 81 mg Acetylsalicylic acid film coated tablet orally once daily with concomitant P2Y12 inhibitor therapy
- Total: Total of all reporting groups
Arm/Group | Apixaban With Acetylsalicylic Acid Film Coated Tablet | Apixaban With Placebo Matching Acetylsalicylic Acid | Vitamin K Antagonist (VKA) With Acetylsalicylic | VKA With Placebo Matching Acetylsalicylic Acid | Total
Number analyzed (Participants) | 1153 | 1153 | 1154 | 1154 | 4614
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.2 (9.12) | 69.3 (9.32) | 70.0 (9.09) | 70.0 (9.13) | 69.9 (9.17)
Age, Customized [Number; unit: Participants]
  < 65 years old | 308 | 333 | 311 | 315 | 1267
  65-80 years old | 664 | 660 | 662 | 657 | 2643
  >=80 | 181 | 160 | 181 | 182 | 704
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 357 | 313 | 339 | 328 | 1337
  Male | 796 | 840 | 815 | 826 | 3277
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 10 | 7 | 5 | 24
  Not Hispanic or Latino | 114 | 123 | 120 | 126 | 483
  Unknown or Not Reported | 1037 | 1020 | 1027 | 1023 | 4107
Race/Ethnicity, Customized [Number; unit: Participants] — Table is for category of Race.
  Participants
    White | 1039 | 1058 | 1043 | 1044 | 4184
    Black/African American | 17 | 12 | 12 | 18 | 59
    Asian | 35 | 35 | 39 | 31 | 140
    American Indian/Alaska Native | 4 | 6 | 2 | 4 | 16
    Native Hawaiian/Other Pacific Islander | 0 | 0 | 0 | 1 | 1
    Other | 47 | 29 | 38 | 43 | 157
    Not Reported | 11 | 13 | 20 | 13 | 57

OUTCOME MEASURES:

1. Primary Outcome: The Rate of International Society on Thrombosis and Haemostasis (ISTH) Major or Clinically Relevant Non-Major (CRNM) Bleeding With Apixaban Versus Vitamin K Antagonist (VKA) During the Treatment Period
Description: Time to first ISTH major or CRNM bleeding during the 6-month period of treatment with Apixaban or VKA.
  N is the number of participants treated with Apixaban or VKA.
  n is the number of participants treated with Apixaban or VKA with major or CRNM bleeding in each treatment group during the 6-month period of treatment.
  Event rates are calculated based on the number of participants with major or CRNM bleeding divided by the sum of the number of days from the first dose of study drug to the event date or censoring date and expressed as percentage per year.
Time Frame: Approximately 6 months
Population: Participants treated with Apixaban or VKA.
  Assessment is only for the Apixaban and VKA interventions.
Measure: Number; unit: Percentage per year
Groups:
- Apixaban: 5 mg or 2.5 mg Apixaban tablets orally twice per day with concomitant P2Y12 inhibitor therapy
- Vitamin K Antagonist: VKA tablets orally once daily with concomitant P2Y12 inhibitor therapy
Arm/Group | Apixaban | Vitamin K Antagonist
Number analyzed (Participants) | 2290 | 2259
Percentage per year | 24.66 | 35.79
Statistical Analysis 1: Comparison: Apixaban vs Vitamin K Antagonist; Separate hierarchical testing was performed for apixaban vs VKA: 1) Non-inferiority for the primary endpoint; Test type: Non-Inferiority — Non-Inferiority (NI) margin = 1.2; p < 0.0001, 1-sided p-value for NI test
Statistical Analysis 2: Comparison: Apixaban vs Vitamin K Antagonist; Separate hierarchical testing was performed for apixaban vs VKA: 2) Superiority for the primary endpoint; Test type: Superiority; p < 0.0001, 2-sided p-value for superiority test; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.58 to 0.82]

2. Primary Outcome: The Rate of ISTH Major or CRNM Bleeding With Aspirin Versus no Aspirin During the Treatment Period
Description: Time to first ISTH major or CRNM bleeding during the treatment period of 6 months with aspirin or placebo.
  N is the number of participants with aspirin or placebo.
  n is the number of participants treated with aspirin or placebo with major or CRNM bleeding in each treatment group during the 6-month period of treatment.
  Event rates are calculated based on the number of participants with event of interest divided by the sum of the number of days from the first dose of study drug to the event date or censoring date and expressed as percentage per year.
Time Frame: Approximately 6 months
Population: Participants treated with aspirin or placebo.
  Assessment is only for the Acetylsalicylic acid film coated tablet or Placebo matching Acetylsalicylic acid film coated tablet interventions.
Measure: Number; unit: Percentage per year
Groups:
- Acetylsalicylic Acid Film Coated Tablet: 81 mg Acetylsalicylic acid film coated tablet orally once daily with concomitant P2Y12 inhibitor therapy
- Placebo Matching Acetylsalicylic Acid Film Coated Tablet: Placebo matching Acetylsalicylic acid film coated tablet orally once daily with concomitant P2Y12 inhibitor therapy
Arm/Group | Acetylsalicylic Acid Film Coated Tablet | Placebo Matching Acetylsalicylic Acid Film Coated Tablet
Number analyzed (Participants) | 2277 | 2279
Percentage per year | 40.51 | 21.03
Statistical Analysis 1: Comparison: Acetylsalicylic Acid Film Coated Tablet vs Placebo Matching Acetylsalicylic Acid Film Coated Tablet; Separate hierarchical testing was performed for aspirin vs placebo: 2) Superiority for the primary endpoint; Test type: Superiority; p < 0.0001, 2-sided p-value for superiority test; Hazard Ratio (HR) = 1.88, 95% CI 2-sided [1.58 to 2.23]

3. Secondary Outcome: Superiority on ISTH Major or CRNM Bleeding for Apixaban Versus VKA
Description: Time to first occurrence during the time the participants were treated with Apixaban or VKA.
  N is the number of participants treated with Apixaban or VKA.
  n is the number of participants treated with Apixaban or VKA with major or CRNM bleeding in each treatment group during the 6-month period of treatment.
  Event rates are calculated based on the number of participants with event of interest divided by the sum of the number of days from the first dose of study drug to the event date or censoring date and expressed as percentage per year.
Time Frame: Approximately 6 months
Population: Participants treated with Apixaban or VKA.
  Assessment is only for the Apixaban or VKA interventions.
Measure: Number; unit: Percentage per year
Arm/Group | Apixaban | Vitamin K Antagonist
Number analyzed (Participants) | 2290 | 2259
Percentage per year | 24.66 | 35.79
Statistical Analysis 1: Comparison: Apixaban vs Vitamin K Antagonist; Separate hierarchical testing was performed for apixaban vs VKA: 2) Superiority for the primary endpoint; Test type: Superiority; p < 0.0001, 2-sided p-value for superiority test

4. Secondary Outcome: The Rate of All-cause Death or All-cause Rehospitalization With Apixaban Versus VKA
Description: Time to first all-cause death or all-cause hospitalization during the during the 6-month treatment period with Apixaban or VKA.
  N is the number of participants treated with Apixaban or VKA.
  n is the number of participants treated with Apixaban or VKA with all-cause death or all-cause hospitalization in each treatment group during the 6-month period of treatment.
  Event rates are calculated based on the number of participants with all-cause death or all-cause hospitalization divided by the sum of the number of days from the first dose of study drug to the event date or censoring date and expressed as percentage per year.
Time Frame: Approximately 6 months
Population: Participants randomized to Apixaban or VKA.
  Assessment is only for the Apixaban or VKA interventions.
Measure: Number; unit: Percentage per year
Arm/Group | Apixaban | Vitamin K Antagonist
Number analyzed (Participants) | 2306 | 2308
Percentage per year | 57.24 | 69.19
Statistical Analysis 1: Comparison: Apixaban vs Vitamin K Antagonist; Separate hierarchical testing was performed for apixaban vs VKA: 3) Superiority for all-cause death and all-cause rehospitalization; Test type: Superiority; p = 0.0033, 2-sided p-value; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.75 to 0.94]

5. Secondary Outcome: The Rate of All-cause Death or All-cause Rehospitalization With Aspirn Versus no Aspirin
Description: Time to first all-cause death or all-cause hospitalization during the 6-month period of treatment with aspirin or placebo.
  N is the number of participants treated with aspirin or placebo.
  n is the number of participants treated with aspirin or placebo with all-cause death or all-cause hospitalization in each treatment group during the 6-month period of treatment.
  Event rates are calculated based on the number of participants with all-cause death or all-cause hospitalization divided by the sum of the number of days from the first dose of study drug to the event date or censoring date and expressed as percentage per year.
Time Frame: Approximately 6 months
Population: Participants randomized to aspirin or placebo.
  Assessment is only for the Acetylsalicylic acid film coated tablet or Placebo matching Acetylsalicylic acid film coated tablet interventions.
Measure: Number; unit: Percentage per year
Arm/Group | Acetylsalicylic Acid Film Coated Tablet | Placebo Matching Acetylsalicylic Acid Film Coated Tablet
Number analyzed (Participants) | 2307 | 2307
Percentage per year | 65.72 | 60.56
Statistical Analysis 1: Comparison: Acetylsalicylic Acid Film Coated Tablet vs Placebo Matching Acetylsalicylic Acid Film Coated Tablet; Separate hierarchical testing was performed for aspirin vs placebo: 3) Superiority for all-cause death and all-cause rehospitalization; Test type: Superiority; p = 0.2219, 2-sided p-value; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.96 to 1.20]

6. Secondary Outcome: The Rate of the Composite Endpoint of Death or Ischemic Events (Stroke, Myocardial Infarction, Stent Thrombosis, Urgent Revascularization) With Apixaban Versus VKA
Description: Time to first occurrence during the 6-month treatment period with Apixaban or VKA.
  N is the number of participants treated with Apixaban or VKA.
  n is the number of participants treated with Apixaban or VKA with death or ischemic events in each treatment group during the during the 6-month period of treatment.
  Event rates are calculated based on the number of participants with death or ischemic events divided by the sum of the number of days from the first dose of study drug to the event date or censoring date and expressed as percentage per year.
Time Frame: Approximately 6 months
Population: Participants randomized to Apixaban or VKA.
  Assessment is only for the Apixaban or VKA interventions.
Measure: Number; unit: Percentage per year
Arm/Group | Apixaban | Vitamin K Antagonist
Number analyzed (Participants) | 2306 | 2308
Percentage per year | 15.85 | 17.17
Statistical Analysis 1: Comparison: Apixaban vs Vitamin K Antagonist; Separate hierarchical testing was performed for apixaban vs VKA: 4) Superiority for all-cause death and ischemic events; Test type: Superiority; p = 0.4370, 2-sided p-value; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.75 to 1.13]

7. Secondary Outcome: The Composite Endpoints of Death and Ischemic Events (Stroke, Myocardial Infarction, Stent Thrombosis, Urgent Revascularization) With Aspirin Versus no Aspirin
Description: Time to first death or ischenic event during the 6-month treatment period with aspirin or placebo.
  N is the number of participants treated with aspirin or placebo.
  n is the number of participants treated with aspirin or placebo with death or ischemic events in each treatment group during the 6-month treatment period.
  Event rates are calculated based on the number of participants with death or ischemic events divided by the sum of the number of days from the first dose of study drug to the event date or censoring date and expressed as percentage per year.
Time Frame: Approximately 6 months
Population: as for outcome 5
Measure: Number; unit: Percentage per year
Arm/Group | Acetylsalicylic Acid Film Coated Tablet | Placebo Matching Acetylsalicylic Acid Film Coated Tablet
Number analyzed (Participants) | 2307 | 2307
Percentage per year | 15.28 | 17.73
Statistical Analysis 1: Comparison: Acetylsalicylic Acid Film Coated Tablet vs Placebo Matching Acetylsalicylic Acid Film Coated Tablet; Separate hierarchical testing was performed for aspirin vs placebo: 4) Superiority for all-cause death and ischemic events; Test type: Superiority; p = 0.1742, 2-sided p-value; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.70 to 1.07]

ADVERSE EVENTS:
Time Frame: Includes adverse events (AEs) with onset on or after the first dose of study medication through 2 days (for non-serious AE) or 30 days (for serious AE) after the last dose of study medication (approximately 7 months).
Description: Note: Within the VKA/placebo arm, 1 participant was enrolled but died prior to dosing and is included only within the All-Cause Mortality table below.
Groups:
- APIXABAN ONLY: Only Apixaban intervention received: 5 mg or 2.5 mg Apixaban tablets orally twice per day
- VKA ONLY: Only VKA intervention received: VKA tablets orally once daily
- ACETYLSALICLIC ACID ONLY: Only acetylsalicylic acid intervention received: 81 mg Acetylsalicylic acid film coated tablet orally once daily
- PLACEBO MATCHING ACETYLSALICLIC ACID ONLY: Only placebo matching acetylsalicylic acid intervention received: placebo matching Acetylsalicylic acid film coated tablet orally once daily
Arm/Group | Apixaban With Acetylsalicylic Acid Film Coated Tablet | Apixaban With Placebo Matching Acetylsalicylic Acid | Vitamin K Antagonist (VKA) With Acetylsalicylic Acid | VKA With Placebo Matching Acetylsalicylic Acid | APIXABAN ONLY | VKA ONLY | ACETYLSALICLIC ACID ONLY | PLACEBO MATCHING ACETYLSALICLIC ACID ONLY
All-Cause Mortality (participants affected / at risk) | 42/1145 | 46/1143 | 38/1123 | 42/1127 | 0/2 | 3/10 | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 53/1145 | 50/1143 | 52/1123 | 55/1126 | 0/2 | 3/10 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 35/1145 | 21/1143 | 33/1123 | 18/1126 | 0/2 | 1/10 | 3/9 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban With Acetylsalicylic Acid Film Coated Tablet (N=1145) | Apixaban With Placebo Matching Acetylsalicylic Acid (N=1143) | Vitamin K Antagonist (VKA) With Acetylsalicylic Acid (N=1123) | VKA With Placebo Matching Acetylsalicylic Acid (N=1126) | APIXABAN ONLY (N=2) | VKA ONLY (N=10) | ACETYLSALICLIC ACID ONLY (N=9) | PLACEBO MATCHING ACETYLSALICLIC ACID ONLY (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 1 | 6 | 3 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 9 | 5 | 3 | 0 | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 4 | 5 | 5 | 2 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac death (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Multimorbidity (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 5 | 3 | 2 | 1 | 0 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Meningoencephalitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 2 | 1 | 3 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 3 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 4 | 0 | 0 | 0 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0 | 5 | 1 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Brain injury (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Shock (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban With Acetylsalicylic Acid Film Coated Tablet (N=1145) | Apixaban With Placebo Matching Acetylsalicylic Acid (N=1143) | Vitamin K Antagonist (VKA) With Acetylsalicylic Acid (N=1123) | VKA With Placebo Matching Acetylsalicylic Acid (N=1126) | APIXABAN ONLY (N=2) | VKA ONLY (N=10) | ACETYLSALICLIC ACID ONLY (N=9) | PLACEBO MATCHING ACETYLSALICLIC ACID ONLY (N=10)
Anaemia (Blood and lymphatic system disorders) | 16 | 3 | 10 | 6 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 8 | 8 | 9 | 5 | 0 | 0 | 1 | 0
Puncture site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 5 | 1 | 2 | 2 | 0 | 0 | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 9 | 3 | 5 | 2 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 3 | 5 | 3 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 4 | 3 | 6 | 1 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT02415400/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT02415400/SAP_001.pdf